CLINICAL TRIAL: NCT03972982
Title: Induction of Long-term Glycemic Remission Via Structured Simplified Short-term Intensive Insulin Therapy in Patients With Newly Diagnosed Type 2 Diabetes: a Multiple Centered, Randomised Controlled Trial.
Brief Title: Effects of Structured Simplified Short-term Intensive Insulin Therapy on Long-term Glycemic Remission
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018YFC1314102
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Newly Diagnosed Type 2 Diabetes; Simplified Short-term Intensive Insulin Therapy; Glycemic Remission

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified regimen group (Experimental): Short-term continuous subcutaneous insulin infusion will be adminstrated to maintained euglycemia for 1 week，Then subsequent therapy using basal insulin plus metformin will be administrated. After withdrawal of the medicine, wearable devices and smart apps will be used for long-term management.
  Interventions: Drug: Simplified intensive insulin therapy regimen
- Routine group (Active Comparator): Inpaitent short-term continuous subcutaneous insulin infusion will be administered to maintained euglycemia for 2 weeks, Then subjects will be follow-up routinely.
  Interventions: Drug: Traditional Short-term Intensive insulin therapy

INTERVENTIONS:
Drug: Simplified intensive insulin therapy regimen — Short-term continuous subcutaneous insulin infusion to maitain near normoglycemica for 1 week, thereafter basal insulin and metformin were subsequently used. Wearable devices and smart apps will be used for lifestyle modification.
  Arms: Simplified regimen group
Drug: Traditional Short-term Intensive insulin therapy — Short-term continuous subcutaneous insulin infusion will be initiate to maitain near normoglycemica for 2 weeks, then patients will be ordinarily follow-up
  Arms: Routine group

SUMMARY:
Short-term intensive insulin therapy is shown to induced glycemic remission, but traditionally patients were hospitalized for 2-4 weeks in order to receive the therapy, the long inpatient period precluded the wide application of the thrapy. This study aims to invesitgate whether simplified regimen is non-inferior to traditional regimen in achieving long-term glycemic remisson.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetes with no prior hypoglycemic agents application, or on hyperglycemic monotherapy for less than 1 week;
* GHbA1c ≥ 9%
* Body mass index between 20-35kg/m2
* Capable to use wearable devices and mobile Apps;
* willling to follow the study protocol and data collection.

Exclusion Criteria:

* Type 1 diabetes or specific types of diabetes;
* Allergic or intolercance to medicine used in the study;
* Acute diabetic complications (diabetic ketoacidosis, hyperosmotic hyperglycemia coma or lactic acidosis);
* Severe diabetic microvascular complications (proliferative retinopathy, clinical proteinuria,uncontrolled diabetic neuropathy and obvious diabetic autonomic neuropathy;
* Glomerular filtration rate less than 50 ml/min
* ALT >2.5 times of the upper limit of normal (ULN), or bilirubin > 1.5 times of ULN；
* Significant Macrovascular disease:acute cerebrovascular accident, acute coronary syndrome or peripheral artery disease that required vascular intervention or amputation 12 months before enrollment;
* Poor blood pressure control (systolic blood pressure≥180mmHg and/or sitting diastolic blood pressure ≥110mmHg) and unable to control under 160/110mmhg within 1 week;
* Hemoglubin level < 100g/L or required regular blood transfusion;
* Chronic cardiac dysfunction with NYHA grade III or above;
* Use of medicines that affect blood glucose for a cumulative time of more than 1 week within the prior 12 weeks, such as oral/venous glucocorticoid, growth hormone, estrogen/ progesterone, high-dose diuretics, antipsychotic drugs. However, low-dose diuretics for antihypertensive purposes (HCTZ < 25mg/d, indapamide < 1.5mg/d) and physiologic replacement of thyroid hormone are allowed;
* Serious systemic disease or malignant tumor, chronic diarrhea, etc；
* Uncontrolled abnormalty in endocrine glands (Cushing's syndrome, hyperthyroidism, etc.);
* Any factors that may affect the participation of the subject in the study or the evaluation of the results；
* Pregnancy or planned pregnancy, lactation subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
remission rate | 24 weeks after withdrawal of the medical intervention
  Remission is defined as fasting plasma glucose less than 7mmol/L and GHbA1c less than 7% without any hypoglycemic agents

CONTACTS AND LOCATIONS:
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China